CLINICAL TRIAL: NCT06920108
Title: TRACE4BUS: Use of the TRACE4BUS Software to Support the Physician in Reporting Breast Ultrasound Results According to the International Classification Standard Breast Image - Reporting and Data System (BI-RADS)
Brief Title: TRACE4BUS for BI-RADS Classification
Status: Not yet recruiting | Type: Observational
Sponsor: DeepTrace Technologies S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: TRACE4BUSv2.0-CIP-1
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; BI-RADS classification; Breast ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort: The investigators propose a retrospective study on patients aged ≥18 years, who have had breast masses detected on ultrasound and considered suspicious for breast cancer by physicians expert in breast ultrasound at the Breast Radiology Unit of the National Cancer Institute, Milan, Italy, from January 1, 2020 to December 31, 2021. These ultrasound images of breast masses will be those acquired in the context of ultrasound-guided core needle biopsy.
- Prospective cohort: The investigators propose a prospective design on consecutive patients (age > 18 years) with breast masses detected by ultrasound and considered suspicious for breast cancer by physicians with experience in breast ultrasound at the same clinic, from the approval data of the Ethics Committee until completion of the expected sample size.

SUMMARY:
The purpose of this clinical study is to evaluate the use of the TRACE4BUS software that is proposed to support the physician in reporting the results of breast ultrasound according to the international classification standard Breast Image - Reporting and Data System (BI-RADS) of the American College of Radiology. This classification is recommended because it reduces the risk of subjective interpretations of descriptive results and prevents these results from being interpreted differently by the physician who evaluated the ultrasound examination, the physician who may have requested the examination, the patient and the patient's trusted physician (family physician or specialist). The BI-RADS classification is based on the evaluation of the shape, size, margins and other characteristics of a possible breast abnormality identified on the ultrasound image by the physician who evaluated the ultrasound examination, characteristics that are not always easy for that physician to evaluate.

The study aims to verify if the BI-RADS classification by the physician can be supported by the TRACE4BUS software. In particular, it refers to the support that the software provides to the physician who has evaluated the ultrasound examination in assigning the BI-RADS category for an abnormality of the breast found to be suspicious by the physician on the basis of qualitative characteristics (shape, size, margins, preferential orientation with respect to the skin plane, internal homogeneity/inhomogeneity, possible acoustic barrier effect, etc.). The TRACE4BUS software, trained on the basis of hundreds of ultrasound images of suspicious breast masses with a certain diagnosis of benignity or malignancy at subsequent diagnostic investigations, performs a quantitative analysis of the ultrasound characteristics of a suspicious breast mass and proposes a BI-RADS category to the physician. In any case, the physician will have complete decision-making power in the final attribution of the BI-RADS category and in the subsequent recommendations or decisions regarding the medical management of the case.

The clinical study also aims to evaluate whether the agreement between physicians in the use of this BI-RADS classification of suspicious breast masses improves with the use of the software.

ELIGIBILITY:
Inclusion Criteria:

1. Retrospective study part:

   * Availability of ultrasound-guided breast biopsy and, in case of B3 lesions at needle biopsy, the vacuum-assisted excision, or surgical specimens or a clinical follow-up outcome in at least 12 months subsequent to the biopsy.
2. Prospective study part:

   * Signed informed consent to participate in the study.

Exclusion Criteria:

1. Retrospective study part:

   * Not availability of ultrasound-guided breast biopsy and, in case of B3 lesions at needle biopsy, the vacuum-assisted excision, or surgical specimens, or a clinical follow-up outcome in at least 12 months subsequent to the biopsy. Age < 18 or > 89 years.
2. Prospective study part:

   * Not availability of Signed informed consent to participate in the study. Age < 18 or > 89 years.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast masses detected at ultrasound imaging and considered suspicious for breast cancer by physicians with experience in breast ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Specificity, positive predictive value, sensitivity and negative predictive value | From enrollment to biopsy up to 12-month follow-up when necessary
  Specificity, positive predictive value, sensitivity and negative predictive value before knowing the BI-RADS category proposed by the TRACE4BUS software and after being informed of the software prediction of BI-RADS category by the TRACE4BUS software.

SECONDARY OUTCOMES:
K-Cohen | 9 months and 18 months
  K-Cohen to measure inter-rater agreement between two physicians before knowing the BI-RADS category proposed by the TRACE4BUS software and after being informed of the software prediction of BI-RADS category by the TRACE4BUS software
Number of correct answers on the use of TRACE4BUS as assessed in the training questionnaire | From date of training in the use of TRACE4BUS software to the physicians to training efficacy questionnaire within 2 weeks
  Number of correct answers in the training questionnaire to measure the effectiveness of the training in the use of TRACE4BUS software after one session. More than 70% (0% minimum score, 100% maximum score) of correct answers are required to demonstrate the effectiveness of the training.
Total scores on the usability of TRACE4BUS as assessed in the usability satisfaction questionnaire | 9 months and 18 months
  Total scores on the usability satisfaction questionnaire to measure the usability satisfaction of TRACE4BUS. More than 70% of satisfaction (0% minimum satisfaction, 100% maximum satisfaction) is required to demonstrate the satisfaction on the usability of TRACE4BUS.

OTHER OUTCOMES:
Number of software deficiencies, adverse software effects and adverse events for participants | 9 months and 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy